CLINICAL TRIAL: NCT07151391
Title: The Use of Guarana to Treat Fatigue in Patients With Neuroendocrine Tumors and Gynecologic Cancers
Brief Title: The Use of Guarana to Treat Fatigue in Patients With Neuroendocrine Tumors and Gynecologic Cancers (Guarana Fatigue)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCI188422
Record Dates: First submitted 2025-08-20; First posted 2025-09-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neuroendocrine Tumors; Gynecologic Cancer
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — guarana powder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guarana (Experimental): The study's goal is to determine the effect of Guarana on symptoms of fatigue
  Interventions: Drug: Guarana
- Placebo (Placebo Comparator): The study's goal is to determine the effect of Guarana on symptoms of fatigue
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guarana — 500 mg oral medication daily
  Other Names: Paullinia cupana
  Arms: Guarana
Drug: Placebo — Oral medication daily
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to learn if the drug guarana improves symptoms of fatigue in patients with neuroendocrine tumors and gynecologic cancers

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years.
* Cohort A (Neuroendocrine Tumor) Only:

  ---Subjects with unresected locally advanced or metastatic well differentiated neuroendocrine tumors who are either on a watch- and-wait approach or receiving treatment with somatostatin analog(s). Patient who received and completed another active treatment but are on a "break" from treatment will be allowed to enroll (e.g., patients that had completed PRRT).
* Cohort B (Gynecological Cancer) Only:

  ---Subjects with early-stage (I or II) ovarian/fallopian-tube cancer in surveillance who have completed all treatment or are receiving adjuvant treatment.
* Or

  ---Subjects with endometrial cancer which is low risk, low-intermediate risk in surveillance, or high-intermediate risk receiving brachytherapy. Risk category is based on GOG criteria.
* ECOG Performance Status ≤ 2.
* Documentation of a score of 4 or higher when answering either of the NCCN-recommended screening questions ("How exhausted do you feel on a scale of 0 to 10?" or "How impaired do you feel by this fatigue on a scale of 0 to 10?") within 4 weeks prior to randomization
* Adequate organ function as defined as:

  * Hematologic:

    * Hemoglobin ≥ 9 g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN) or ≤3 x ULN with documented liver involvement and/or Gilbert's disease
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN ----Subjects with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
  * Renal:

    ---Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula
  * For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women < 50 years of age:

      ----Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or

      ----Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥ 50 years of age:

      * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments and luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or Amenorrhea for 24 months following cessation of all exogenous hormonal treatments, if applicable; or
      * Had radiation-induced menopause with last menses >1 year ago; or
      * Had chemotherapy-induced menopause with last menses >1 year ago; or
      * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
  * Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception.
  * Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* For the Neuroendocrine Tumor cohort: Receiving treatment with Cytotoxic Chemotherapy, Radiation Therapy, PRRT or TKIs within 6 weeks prior to the first dose of study treatment.
* For the Gynecological Cancer cohort: Receiving any systemic treatment besides those listed in Inclusion 3-Cohort B (Gyn only) within 6 weeks prior to the first dose of study treatment.
* Untreated or uncontrolled endocrinopathy which is likely to significantly impact study participation.
* History of significant autoimmune disease in the opinion of the investigator that is likely to significantly impact study participation.
* Prior use of guarana supplements within two months of consent.
* Self-reported "caffeine sensitivity" defined as excessive unwanted feelings of anxiousness, jitteriness, difficulty sleeping, or anxiety after caffeine exposure, which in the opinion of the Investigator is likely to negatively impact study participation.
* Concurrent use of psychostimulants (e.g., lisdexamfetamine, methylphenidate).
* Major surgery within 4 weeks prior to starting study therapy or subjects who have not fully recovered from major surgery.
* The diagnosis of another malignancy which, in the opinion of the investigator, is likely to negatively impact subject safety or study aims.
* Known brain metastases or cranial epidural disease.

  --Note: Subjects with brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the first dose of study treatment.
* Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

  --Cardiovascular disorders:
  * Significant symptomatic carcinoid heart disease in the opinion of the investigator
  * Congestive heart failure New York Heart Association Class III or IV, unstable angina pectoris, serious cardiac arrhythmias.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events) within 3 months before the first dose.
  * Thromboembolic events (eg, deep venous thrombosis, pulmonary embolism) within 1 month before the first dose.
  * QTc prolongation defined as a QTcF > 500 ms.
  * Known congenital long QT.
  * Uncontrolled hypertension per investigator assessment or grade 3 hypertension per CTCAE v.5.0
  * Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the therapy through a feeding tube], social/ psychological issues, etc.)
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

  --Note: Subjects on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Known active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known hypersensitivity or allergy to investigational product (IP).
* Subjects taking prohibited medications as described in Section 6.6.2 or medications for which caffeine intake is contraindicated including: β-adrenergic agonists, and/or medications that contain pseudoephedrine. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Stage 1 Primary Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Fatigue 12 (EORTC QLQ-FA12) questionnaire scores from screening to Day 21 of guarana treatment. | up to 21 days after initiation of study intervention
  To assess the use of guarana to improve symptoms of fatigue in patients with NETs and Gynecologic (Ovarian/Fallopian Tube and Endometrial) cancers and to estimate the Cohen's effect size for planning of the randomized controlled trial in stage II.
  This outcome measure will report 3 sub-scales (Physical Fatigue Score, Emotional Fatigue Score, and Cognitive Fatigue Score) and two single-item measures (Interference with daily life and Social sequelae score).
  All of the scales and single-item measures range in score from 0 to 100. For all the scales and single items, a high score represents a high level of symptomatology or problems.
Stage 2 Change in EORTC QLQ-FA12 questionnaire scores from screening to days 21 and 42 of treatment. | up to 42 days after initiation of study intervention
  To evaluate if the EORTC QLQ-FA12 score changes from baseline to Day 21 and 42 days differs between the guarana treated arm and the placebo arm.
  This outcome measure will report 3 sub-scales (Physical Fatigue Score, Emotional Fatigue Score, and Cognitive Fatigue Score) and two single-item measures (Interference with daily life and Social sequelae score).
  All of the scales and single-item measures range in score from 0 to 100. For all the scales and single items, a high score represents a high level of symptomatology or problems.

SECONDARY OUTCOMES:
The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment. | up to 5 week after initiation of study intervention
  To assess the safety and tolerability of guarana in the study population.
Quality of Life (QoL) - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Gastrointestinal Neuroendocrine Tumors (EORTC QLQ-GINET21) | up to 5 week after initiation of study intervention
  This outcome measure will report the sub-scales and single-item measures of the EORTC QLQ-C21NET for patients in the endometrial cohort
  EORTC QLQ-C21NET will report 5 sub-scales (Endocrine, Gastrointestinal, Treatment-Related, Disease-Related Worries, Social Functioning) and 5 single-item measures (Weight Loss, Weight Gain, Muscle and/or Bone Pain, Information, Sexual Functioning)
  All of scales and single-item measures range in score from 0 to 100. For all the scales and single items, a high score represents a high level of symptomatology or problems.
Quality of Life (QoL) - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Endometrial Cancer Module 24 (EORTC QLQ-EN24) | up to 5 week after initiation of study intervention
  This outcome measure will report the sub-scales and single-item measures of the EORTC QLQ-EN24 for patients in the endometrial cohort
  EORTC QLQ-EN24 will report 7 sub-scales (Lymphoedema, Urological, Gastrointestinal, Poor body image, Sexual/vaginal problems, Tingling/numbness, Muscular pain) and 6 single-item measures (Sexual interest, Sexual activity, Sexual enjoyment, Pain in back and pelvis, Hair loss, Taste change)
  All of the scales and single-item measures range in score from 0 to 100. For all the scales and single items, a high score represents a high level of symptomatology or problems.
Quality of Life (QoL) - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Ovarian Cancer 28 (EORTC QLQ-OV28) | up to 5 week after initiation of study intervention
  This outcome measure will report the sub-scales and single-item measures of the EORTC QLQ-OV28 for patients in the ovarian/fallopian tube cohort.
  EORTC QLQ-OV28 reports 8 sub-scales (Abdominal/GI Scale, Peripheral Neuropathy, Hormonal, Body image, Attitude to disease/treatment, Hair Loss, Chemotherapy side effects, Sexuality) and 2 single-item measures (Indigestion or Heartburn, Taste)
  All of the scales and single-item measures range in score from 0 to 100. For all the scales and single items, a high score represents a high level of symptomatology or problems.
Subjective patient experience with guarana supplementation | up to 5 week after initiation of study intervention
  This outcome will assess the subjective experience of participants with guarana supplementation. At the end of the study, participants will be asked: "How would you describe your experience with guarana supplementation?". Responses will be recorded using a three-point Likert scale (Positive, Neither positive or negative, or Negative).
  This outcome measure will report the count of participants selecting each response category.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States